CLINICAL TRIAL: NCT02711111
Title: Effect of Bone-anchored Protraction on Maxillary Growth in the Young Child
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Joeri Meyns, J. Meyns, M.D., D.M.D., oral and maxillofacial Surgery, principal investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKA Genk
Record Dates: First submitted 2016-03-07; First posted 2016-03-17 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Maxillary Hypoplasia; Malocclusion, Angle Class III
MeSH Terms: conditions — Retrognathia; Malocclusion, Angle Class III | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- orthodontic bone anchor (Experimental): new bone anchor device, which creates anterior traction on the upper jaw. Placed on the chin-region intra-orally.
  Interventions: Device: orthodontic bone anchor
- face mask protraction (Active Comparator): control group, conventional treatment method. Face mask creates anterior traction on the upper jaw
  Interventions: Device: Face mask

INTERVENTIONS:
Device: Face mask — to apply for on the upper jaw (12 - 14 hrs / day) via extra-oral elastics to the face mask
  Other Names: face mask of dealer
  Arms: face mask protraction
Device: orthodontic bone anchor — to apply force on the upper jaw (24 / 7) via intra-oral elastics on the bone-anchor
  Other Names: mentoplate, PSM medical solutions, Tuttlingen, Germany
  Arms: orthodontic bone anchor

SUMMARY:
Class III malocclusions may originate in a retrognathic maxilla, a prognathic mandible or both. Young patients with class III malocclusion and maxillary hypoplasia are conventionally treated with a protraction facemask in order to stimulate forward growth of the upper jaw. This treatment option is often inducing unwanted side effects including mesial migration of the teeth in the upper jaw and clockwise rotation of the mandible. Because skeletal effects are often difficult to achieve with this approach, more pronounced class III malocclusions cannot be addressed by face mask therapy. These children cannot be treated during childhood and end up in major orthognathic surgery at full-grown age. To be able to treat also the more pronounced class III malocclusion and to minimize dentoalveolar compensations new treatment methods were developed which uses skeletal anchorage.

DETAILED DESCRIPTION:
Rationale:

Class III malocclusions may originate in a retrognathic maxilla, a prognathic mandible or both. Young patients with class III malocclusion and maxillary hypoplasia are conventionally treated with a protraction facemask or reverse twin block appliance in order to stimulate forward growth of the upper jaw. This treatment option is often inducing unwanted side effects including mesial migration of the teeth in the upper jaw and clockwise rotation of the mandible. Because skeletal effects are often difficult to achieve with this approach, more pronounced class III malocclusions cannot be addressed by face mask therapy. These children cannot be treated during childhood and end up in major orthognathic surgery at full-grown age.

To be able to treat also the more pronounced class III malocclusion and to minimize dentoalveolar compensations new treatment methods were developed which uses skeletal anchorage. In maxillary deficiency cases it's common to have the deficiency anteroposteriorly as well as transversely. Opening of the midpalatal suture by rapid expansion can correct the transverse hypoplasia and may produce more anterior movement of the maxilla. The proposed technique enables to start skeletal anchorage treatment at an earlier age, which also has the potential of more growth modification during treatment.

Objective:

To compare a new technique of skeletal traction with incorporation of maxillary expansion to conventional treatment protocols.

Study design:

This is a RCT

Study population:

Healthy human volunteers (7- 14 yrs old) with class III malocclusion due to maxillary deficiency.

Intervention:

The intervention consists of the application of a mentoplate (anchored with screws to the bone) in the lower jaw and two screws in the upper jaw (palate). Expansion in the upper jaw is achieved by a classic Hyrax appliance, connected to these screws. Anterior movement of the maxilla is subsequently accomplished by intermaxillary elastic traction to the mentoplate.

Control group (conventional treatment):

Anterior movement of the maxilla accomplished by elastic traction to a face mask

Main study parameters/endpoints:

The main study parameter is the difference in the amount of forward growth of the upper jaw and mid-face (measured with a cone beam CT) compared to the growth that is observed with conventional treatment.

A cone beam CT will be made before the start of traction therapy (baseline) and after 1 year of therapy to evaluate the amount of expansion and forward growth of the maxilla.

One last cone beam CT will be produced at the end of growth, 5 years after start of the orthodontic traction, to evaluate the long-term stability of the obtained advancement.

Other end-points will be patients' satisfaction and complication-rate.

ELIGIBILITY:
Inclusion Criteria:

healthy subjects 7 - 14 years old Class III occlusion maxillary hypoplasia good oral hygiene no craniofacial syndrome

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
effect of bone-anchored protraction on maxillary growth in the young child, 1 year with 3D analysis | 1 year
  assessment of anterior growth of the upper jaw, 1 year after start of treatment
effect of bone-anchored protraction on maxillary growth in the young child, 5 years, with 3D analysis | 5 years
  assessment of anterior growth of the upper jaw, 5 years after start of treatment

SECONDARY OUTCOMES:
complications registration | 1 year
  registration of complications due to the use of the new orthodontic bone anchor (mentoplate)
patient satisfaction | 1 year
  registration of the patient satisfaction, easy to use

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Belgium

REFERENCES:
- [Derived] Meyns J, Meewis J, Dons F, Schreurs A, Aerts J, Shujaat S, Politis C, Jacobs R. Long-term comparison of maxillary protraction with hybrid hyrax-facemask vs. hybrid hyrax-mentoplate protocols using Alt-RAMEC: a 5-year randomized controlled trial. Eur J Orthod. 2025 Feb 7;47(2):cjaf011. doi: 10.1093/ejo/cjaf011. PMID 40105065